CLINICAL TRIAL: NCT00427492
Title: Effect of Postoperative Laxative on Bowel Function After Colonic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Jens Andersen. Consultant Surgeon, Copenhagen University Hospital - Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 02 290964
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Colonic Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesia (Active Comparator): Medical laxative
  Interventions: Drug: Magnesia; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesia — Tablet magnesia 500mg. 2 tablet 2 times a day for a week
  Arms: Magnesia
Drug: Placebo

SUMMARY:
Randomised doublet blinded study of the effect of tablet Magnesia (laxative) on post operative bowel ileus after open colonic resection. Material: 56 patients in two equal groups. Primary endpoint: Bowel function. Secondary endpoints: Intake of food and drinks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned elective colonic resection

Exclusion Criteria:

* Previous extended abdominal surgery
* Pregnancy
* Opioid or alcohol abuse

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time to defecation after colonic resection | 2-8 days

CONTACTS AND LOCATIONS:
Overall Officials: Jens Andersen, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University hospital Hvidovre, Hvidovre, Denmark